CLINICAL TRIAL: NCT00411294
Title: The Effect of Ergocalciferol Treatment on 25-Hydroxyvitamin D Levels and Plasma Intact PTH in Patients With Chronic Kidney Disease Stage 3 and 4
Brief Title: Ergocalciferol in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Saint Louis VA Medical Center (U.S. Federal Agency)
Other Study IDs: ZA-01
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2006-12-13 (Estimated); Status verified 2006-12

CONDITIONS: Chronic Kidney Disease
Keywords: ergocalciferol; chronic kidney disease; secondary hyperparathyroidism; vitamin D deficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
To examine the effect of ergocalciferol treatment on 25-hydroxyvitamin D and PTH levels in patients with CKD stage 3 and 4

ELIGIBILITY:
Inclusion Criteria:

* Patient with CKD stage 3 or 4 whose 25-hydroxyvitamin D levels are below 30 ng/ml and plasma intact PTH levels >70 pg/ml.

Exclusion Criteria:

* Patients who are on any form of active vitamin treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ziyad Al-Aly, M.D., Principal Investigator — VAMC-Saint Louis
Locations (1):
- Saint Louis VA Medical Center, St Louis, Missouri, United States

REFERENCES:
- [Derived] Al-Aly Z, Qazi RA, Gonzalez EA, Zeringue A, Martin KJ. Changes in serum 25-hydroxyvitamin D and plasma intact PTH levels following treatment with ergocalciferol in patients with CKD. Am J Kidney Dis. 2007 Jul;50(1):59-68. doi: 10.1053/j.ajkd.2007.04.010. PMID 17591525